CLINICAL TRIAL: NCT06271811
Title: Evaluating the Impact of Flossing Band Integration in Conventional Physiotherapy for Patellofemoral Pain Syndrome
Brief Title: Flossing Band Integration in Conventional Physiotherapy for Patellofemoral Pain Syndrome
Acronym: flossing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: University of Jaen (Unknown)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJAPFPS
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Anterior Knee Pain Syndrome; Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; physiotherapy; mind-body; flossing band
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The intervention protocol is centered on neuromuscular training, targeting the strengthening of key muscle groups including the quadriceps, hamstrings, and hip abductors, which are vital for knee stabilization. This approach is supported by previous research, emphasizing the importance of these muscle groups in knee joint health. Complementing this, proprioceptive exercises, such as single-leg balances and controlled knee bends, were incorporated to enhance joint position sense, aligning with the guidelines set forth by Powers et al., 2010.
  The intensity of these exercises is progressively increased, tailored to each patient's tolerance and improvement. The protocol stipulates two sessions per week over eight weeks.
  Interventions: Other: Conventional physiotherapy
- Intervention group (Experimental): The application of flossing to the knee commences with a preliminary evaluation of the joint range of motion and pain perception. The band is wrapped around the knee, starting with an approximate tension of 50% for the first wrap and escalating to a tension of 60-80% in subsequent wraps. It is essential to overlap the band with each wrap, moving from a distal to the proximal direction (bottom to top), which aids in enhancing drainage. Continuous monitoring of the patient is critical to ensure that excessive pressure is not being applied. This can be achieved by palpating the pulse on the dorsum of the foot or inner ankle, and observing if the skin regains its normal color after pressing the area with fingers. Should the patient experience strong tingling or pain, the bandage must be immediately removed. The duration of the band's application varies between 2 to 5 minutes, depending on patient tolerance, a methodology informed by existing research.
  Interventions: Procedure: Flossing band

INTERVENTIONS:
Procedure: Flossing band — The application of flossing to the knee commences with a preliminary evaluation of the joint range of motion and pain perception. The band is wrapped around the knee, starting with an approximate tension of 50% for the first wrap and escalating to a tension of 60-80% in subsequent wraps. It's essential to overlap the band with each wrap, moving from a distal to the proximal direction (bottom to top), which aids in enhancing drainage. Continuous monitoring of the patient is critical to ensure that excessive pressure is not being applied. This can be achieved by palpating the pulse on the dorsum of the foot or inner ankle, and observing if the skin regains its normal color after pressing the area with fingers. Should the patient experience strong tingling or pain, the bandage must be immediately removed. The duration of the band's application varies between 2 to 5 minutes, depending on patient tolerance, a methodology informed by existing research.
  Arms: Intervention group
Other: Conventional physiotherapy — The intervention protocol is centered on neuromuscular training, targeting the strengthening of key muscle groups including the quadriceps, hamstrings, and hip abductors, which are vital for knee stabilization. This approach is supported by previous research, emphasizing the importance of these muscle groups in knee joint health. Complementing this, proprioceptive exercises, such as single-leg balances and controlled knee bends, were incorporated to enhance joint position sense, aligning with the guidelines set forth by Powers et al., 2010.
  The intensity of these exercises is progressively increased, tailored to each patient's tolerance and improvement. The protocol stipulates two sessions per week over eight weeks.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to assess the efficacy of adding flossing band therapy to conventional physiotherapy in patients diagnosed with Patellofemoral Pain Syndrome (PFPS). The main questions it aims to answer are:

* Does combining flossing band therapy with conventional physiotherapy lead to greater improvements in pain, strength, and function compared to conventional physiotherapy alone?
* What are the effects of flossing band therapy on knee functionality and muscle strength in PFPS patients? Participants will be randomly assigned to either the Standard Physiotherapy group or the Flossing Band and Physiotherapy group. In addition to conventional physiotherapy, participants in the Flossing Band group will undergo sessions where a flossing band is applied around the knee joint to provide moderate compression. Researchers will compare the two groups to determine if the addition of flossing band therapy enhances treatment outcomes for PFPS.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the efficacy of integrating flossing band therapy into conventional physiotherapy for individuals diagnosed with Patellofemoral Pain Syndrome (PFPS). A double-blinded, randomized controlled trial was conducted to evaluate the influence of adding flossing band application to conventional physiotherapy based on 8 weeks of resistance training in patients with PFPS. The study was approved by the research ethics committee of the University of Jaén and conducted in accordance with the Code of Ethics of the World Medical Association for human studies (Declaration of Helsinki). A sample of 50 participants diagnosed with PFPS were randomly allocated into two distinct groups: the Standard Physiotherapy Group (SPG) and the Flossing Band and Physiotherapy Group (FBPG). Eligibility criteria included a clinical diagnosis of PFPS, retro patellar pain for at least three months, and no recent medical treatment or lower extremity surgery within the last six months. Participants underwent assessments at baseline and after 8 weeks of rehabilitation protocols, including standardized measures of pain intensity, knee functionality, and overall mobility. The intervention protocols involved either conventional physiotherapy focused on neuromuscular training or a combined treatment regimen of conventional physiotherapy along with additional flossing band therapy targeting the knee region. Researchers applied rigorous blinding protocols to ensure impartial evaluations and minimize bias. Outcome measures included the Kujala Anterior Knee Pain Scale (AKPS), handheld dynamometry for knee extensor muscle strength, a visual analog scale (VAS) for pain assessment, and the Lower Extremity Functional Scale (LEFS) for self-reported function, isokinetic variables, including peak torque, total work, and average power, were assessed using the Biodex System 4 dynamometer and emotional and psychological variables. The study aimed to determine if the addition of flossing band therapy enhances treatment outcomes for PFPS compared to conventional physiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Patellofemoral Pain Syndrome or patellofemoral misalignment, as confirmed by clinical signs and/or imaging studies (e.g., knee CT scans).
* An age range of 18 to 50 years, to include a broad spectrum of the population affected by PFPS.
* Experience retro patellar pain for at least three months, including pain at rest or during activities such as ascending or descending stairs, jumping, running, squatting, kneeling, or prolonged sitting.
* Pain or apprehension upon mobilization of the patella, and/or crepitus accompanied by pain during activities like squats.
* No history of medical treatment, physiotherapy specifically targeting PFPS, or lower extremity surgery within the last six months.

Exclusion Criteria:

* A history of significant lower extremity, pelvic, or spinal surgery/fracture, or traumatic lesions of ligaments or meniscus within the past six months.

  * Presence of other orthopedic conditions (e.g., ligament rupture, meniscal tears), neurological disorders (e.g., multiple sclerosis, paralysis), rheumatological diseases (e.g., rheumatoid arthritis, ankylosing spondylitis), or congenital conditions leading to osteoarthrosis.
  * Current pregnancy.
  * A history of connective tissue disease, patellofemoral dislocation or subluxation, or osteoarthrosis of the knees.
  * Use of sedatives or muscle relaxants that may alter muscle tone.
  * Other forms of anterior knee pain (e.g., Osgood-Schlatter disease, tendon pain, bursitis).
  * A history of referred pain from the lumbar spine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Disability related to patellofemoral pain | From baseline to 8 weeks
  The Kujala Anterior Knee Pain Scale was employed to assess this variable. is a well-established tool used to evaluate symptoms and functional limitations in individuals with patellofemoral pain syndrome. This self-reported questionnaire comprises 13 items, each rated to provide a total score ranging from 0 to 100, where higher scores denote better knee function and fewer symptoms. While specific cut-off points are not universally defined, scores closer to 100 generally indicate minimal patellofemoral issues.
Knee extensor muscle strength | From baseline to 8 weeks
  In addition to isokinetic variables assessed with the Biodex System 4 dynamometer, manual handheld dynamometry was employed to measure knee extensor muscle strength, providing a comprehensive evaluation of muscle function in individuals with Patellofemoral Pain Syndrome.
Pain report | From baseline to 8 weeks
  Pain was measured using a visual analogue scale (VAS). The VAS consists of a 10-cm line, with the left extremity representing (the absence of pain) and the right extremity indicating (the worse pain devisable). Participants were asked to indicate on the scale their current level of pain being higher values related to more intense pain.

SECONDARY OUTCOMES:
Self-reported function | From baseline to 8 weeks
  Self-reported function: The lower limb function was assessed by the Lower Extremity Functional Scale (LEFS) is a valid and reliable instrument to determine the functional status of acute and chronic lower extremity musculoskeletal dysfunction. It is a 20-item questionnaire whose items are ranged in a five-point scale ranging from zero to four to assess the difficulty in performing different tasks due to physical dysfunction in the lower extremities. The final score of all the items is calculated on a 0-80 score scale, correlated with low and high functional levels respectively, and has been deemed to be a valid and reliable self-reported assessment tool
Short Form-36 (SF-36) | From baseline to 8 weeks
  The SF-36 is widely utilized as a comprehensive measure of health-related quality of life. It comprises 36 items categorized into eight domains: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health. Additionally, it offers summary scores for the physical and mental components (PCS and MCS), with higher scores indicating better overall health-related quality of life.
Berg Balance Scale (BBS) | From baseline to 8 weeks
  This assessment tool is employed for balance evaluation. It comprises 14 items, each rated from 0 to 4, with the scores aggregated to yield a total score ranging from 0 to 56. A higher total score signifies improved balance. Scores between 0 and 20 indicate wheelchair mobility, 21 to 40 suggest walking with assistance, while a score of 41 to 56 indicates independent walking ability.
Pittsburgh Sleep Quality Index | From baseline to 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire used to assess sleep quality and disturbances over a one-month time interval. It evaluates seven components of sleep, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. Each component is scored on a scale of 0 to 3, with higher scores indicating poorer sleep quality. The total score, which ranges from 0 to 21, is calculated by summing the scores of the seven components, with higher scores indicating worse overall sleep quality. The PSQI is widely used in both clinical and research settings to evaluate sleep patterns and disturbances.
Brief Pain Questionnaire | From baseline to 8 weeks
  The Brief Pain Inventory (BPI) is a widely used self-report questionnaire designed to assess the severity of pain and its impact on various aspects of daily functioning. It consists of two main sections: the Pain Severity Scale and the Pain Interference Scale. The Pain Severity Scale assesses the intensity of pain at its "worst," "least," "average," and "right now" over the past week, rated on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). The Pain Interference Scale evaluates the degree to which pain interferes with various domains of daily life, such as general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. Responses are also rated on a scale from 0 (does not interfere) to 10 (completely interferes).
Perceived Stress Scale | From baseline to 8 weeks
  The Perceived Stress Scale (PSS) is a self-report questionnaire designed to measure the perception of stress in individuals over the past month. It consists of 10 items that assess the degree to which situations in one's life are appraised as stressful. Respondents rate the frequency of their feelings and thoughts related to stress on a scale from 0 (never) to 4 (very often). The items cover various aspects of stress, including feelings of unpredictability, lack of control, and overwhelm. The scores for each item are summed to obtain a total score, with higher scores indicating higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: David Cruz Diaz, PhD, Study Director — University of Jaén
Locations (1):
- University of Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No